CLINICAL TRIAL: NCT03829670
Title: The Impact of Cytochrome P450 Abnormalities in Patients With Delirium. A Pilot Study.
Brief Title: The Impact of Cytochrome P450 Abnormalities in Patients With Delirium.
Status: Completed | Type: Observational
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: AHC IRB 6915
Record Dates: First submitted 2019-02-01; First posted 2019-02-04 (Actual); Last update posted 2024-10-04 (Actual); Status verified 2024-09

CONDITIONS: Delirium, Cytochrome P-450 Enzyme System
MeSH Terms: conditions — Delirium

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — One pink (K2EDTA) 6.0 mL (also acceptable: light blue (3.2% sodium citrate) 2.7 mL)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Delirium Group: 1. UBACC: University of California, San Diego Brief Assessment of Capacity to Consent.
  2. The participant may decline participation after this UBACC (University of California, San Diego Brief Assessment of Capacity to Consent) assessment and will be removed from the study.
  3. The Short IQCODE (Informant Questionnaire on Cognitive Decline in the Elderly) is administered to the legally authorized representative or caregiver by Dr. Schmidt. If the potential participant scores 3.3 or lower, the participant will continue in the delirium group. If higher, patient likely with pre-existing dementia. These patients are not eligible for study participation.
  4. Delirium Rating Scale 98 will be performed on the ALGH (Advocate Lutheran General Hospital) rehabilitation unit
  5. Cytochrome P450 testing
  6. Delirium Status: Admission, Hospital Discharge, Outpatient Visit
  7. FIM (The Functional Independence Measure) scores on admission and discharge. FIM efficiency score.
  Interventions: Diagnostic Test: Cytochrome P450 test
- Patients without delirium: 1. Cytochrome P450 testing
  2. Delirium Status: Admission, Hospital Discharge, Outpatient Visit
  3. FIM (The Functional Independence Measure) scores on admission and discharge. FIM efficiency score.
  Interventions: Diagnostic Test: Cytochrome P450 test

INTERVENTIONS:
Diagnostic Test: Cytochrome P450 test — Blood samples will be drawn for cytochrome P450 testing.
  Other Names: CYP2D6, CYP2C9, CYP2C19

SUMMARY:
Objectives:

1. To examine whether patients with delirium have higher prevalence of cytochrome-P450 abnormalities compared to patients without delirium.
2. To examine whether the severity of delirium is related to a specific cytochrome P450 genotype.
3. To examine the persistence of delirium at 6-8 weeks stratified by presence of cytochrome p450 abnormalities
4. To examine whether delirium persistence is impacted by types of medications administered during their hospital stay.

DETAILED DESCRIPTION:
Delirium is a costly and devastating illness affecting older patients in the hospital. Its prevalence increases as patients get older and sicker. There is scientific evidence that delirium affects cognitive function for a prolonged period of time and in many cases irreversibly. The economic burden on health care and emotional burden on the caregivers of patients with delirium is tremendous. We think that our study may contribute to developing prevention strategies for delirium in the hospital. We propose genetic testing of older patients to determine their ability to metabolize commonly used medications in the hospital. This will give medical professionals and pharmacists an ability to adjust dosages of medications based on the patient's genetic profile.

ELIGIBILITY:
Inclusion Criteria:

1. Patients age 18 and older admitted to the ALGH (Advocate Lutheran General Hospital) rehabilitation unit
2. One or more of the Following Principle Diagnosis:

   Principle stroke diagnosis Principle Cardiac-Post cardiac surgery Principle Spinal surgery
3. Non-English speakers are not anticipated. However, there is an available interpreter services already on the unit and this interpreter's services will be utilized. https://www.languageline.com/ However, we will utilize that AHC IRB approved short forms if a potential subject presents itself.

Exclusion Criteria:

1. Stroke patients with any diagnosed aphasia
2. Spinal surgery, as a result of trauma
3. Pregnant women
4. Prisoners
5. Patients with dementia (score of greater than 3.3 on short IQCODE questionnaire) (Long Term Cognitive Impairment after Critical Illness, NEJM, 2013, Pandharipande et al.)
6. Patients with cirrhosis and liver failure
7. Patients with renal failure requiring dialysis
8. Recent blood transfusion

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to the Rehabilitation Unit at Lutheran General Hospital will be approached to participate in this case-control study. Patients will be assigned to the case group once identified with delirium by the Psychology staff. Control group will consist of patients without delirium upon assessment by the Psychology staff. The Delirious patients will then be matched to a control patient hospitalized in the Rehabilitation Lutheran General Unit.
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2019-01-31 (Actual); Primary Completion 2020-06-24 (Actual); Study Completion 2020-06-24 (Actual)

PRIMARY OUTCOMES:
• Rates of cytochrome P450 in cases (delirium patients) compared to controls (non-delirium patients). | 2 years
  Statistical Analysis Plan: Descriptive statistics will be presented as mean ± SD for continuous variables and percentage/count for dichotomous/categorical variables. Chi-square test and t-test will be used to compare distribution of variables of interest between the two groups. Logistic regression analysis will be performed to estimate the risk of PEP while adjusting for all potential confounding factors.

CONTACTS AND LOCATIONS:
Overall Officials: David Ronin, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Advocate Health Care, Park Ridge, Illinois, United States

IPD SHARING:
Plan to Share IPD: No
We will de-identify the data once the study is completed.

REFERENCES:
- See also: Pinto, N., & Dolan, M. E. (2011). Clinically relevant genetic variations in drug metabolizing enzymes. Current Drug Metabolism, 12(5), 487-97. — https://doi.org/10.2174/138920011795495321
- See also: Maldonado, J. R. (2008). Delirium in the Acute Care Setting: Characteristics, Diagnosis and Treatment. Critical Care Clinics. — https://doi.org/10.1016/j.ccc.2008.05.008